CLINICAL TRIAL: NCT06107855
Title: Comparison of Low-dose Maximal-intent Versus Controlled-tempo Resistance Training on Quality-of-life, Functional Capacity, and Strength in Untrained Healthy Adults: a Randomised Controlled Trial
Brief Title: Low-dose Maximal-intent Versus Controlled-tempo Resistance Training on Quality-of-life in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45459
Record Dates: First submitted 2023-09-18; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Quality of Life
Keywords: Activities of Daily Living; Balance; Independence; Mobility; Untrained

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal-intent Resistance Training (Experimental): The MI group was instructed and encouraged to deliberately commit to exerting maximal effort and force during the concentric phase of the leg press with the intention of achieving the greatest velocity possible.
  Interventions: Other: Leg Press Resistance Training Machine
- Controlled-tempo Resistance Training (Experimental): While the CT group followed the metronome for both eccentric and concentric phases.
  Interventions: Other: Leg Press Resistance Training Machine

INTERVENTIONS:
Other: Leg Press Resistance Training Machine — Participants used said unilateral leg press at 60% one-repetition max for either 3 sets x 5 reps, or 5 sets x 5 reps, at either maximal- or controlled-tempo-intent.

SUMMARY:
The aims of this study were to:

1. Compare the effects of low-dose Maximal Intent and Controlled Tempo Resistance Training on untrained healthy adults' quality-of-life, functional capacity, and strength.
2. Qualitatively explore perceptions of Maximal Intent and Controlled Tempo Resistance Training.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were between 30-60 years old
* Uninjured
* Had no cardiovascular or neuromuscular conditions
* Had not participated in lower-limb RT in the previous six months.

Exclusion Criteria:

* Participants were excluded if they had either taken part in any lower-limb RT in the last six months
* Had underlying health condition(s) that prevented them from participating in RT
* Regularly met or exceeded the UK recommended PA guideline of 150-minutes of moderate to intense PA per week.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Quality-of-life | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Participant quality of life (focus group questions & SF-36)

SECONDARY OUTCOMES:
Balance | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Using the biodex SD to do a 3 x 20s double-foot eyes-open balance test on Level 6.
6-minute Walk Test (6MWT) | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  a "brisk"-paced 6-minute walk test.
Timed-up-and-go (TUG) | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Standing from a chair, walking to a point 3 metres away, turn, and return to the chair as quick as possible whilst walking.
30-second sit-to-stand (30s-STS) | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Maximal amount of repetitions a participant can stand up from a chair in 30-seconds.
Strength (1RM) | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Participants one-repetition max on leg press
BMI | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Additional measures calculated from participants test results
Strength-to-mass | The time frame for my testing intervals will be conducted at specific time points: at baseline, Week 1, Week 4, and Week 9, out of a total study duration of 9 weeks.
  Additional measures calculated from participants test results

CONTACTS AND LOCATIONS:
Overall Officials: Gill Barry, PhD, Principal Investigator — Northumbria University
Locations (1):
- Nortuhmbria University, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson LT, Behm DG, Goodall S, Mason R, Stuart S, Barry G. Effects of maximal-versus submaximal-intent resistance training on functional capacity and strength in community-dwelling older adults: a systematic review and meta-analysis. BMC Sports Sci Med Rehabil. 2022 Jul 16;14(1):129. doi: 10.1186/s13102-022-00526-x. PMID 35842655
- [Derived] Pearson LT, Fox KT, Keenan A, Behm DG, Stuart S, Goodall S, Barry G. Comparison of low-dose maximal-intent versus controlled-tempo resistance training on quality-of-life, functional capacity, and strength in untrained healthy adults: a comparative effectiveness study. BMC Sports Sci Med Rehabil. 2024 Mar 23;16(1):72. doi: 10.1186/s13102-024-00847-z. PMID 38521946